CLINICAL TRIAL: NCT05715515
Title: Clinical Evaluation of the Panbio™ COVID-19/Flu A&B Rapid Panel Professional Use Device and the Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDRD-H-029-P
Record Dates: First submitted 2023-01-09; First posted 2023-02-08 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Influenza A; Influenza Type B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal sampling/Testing (Self-Test) + Nasopharyngeal sampling/Testing (Professional Use) (Experimental): Lay users (self-tester or caregiver) will be provided with a Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test kit. Each lay user will collect one mid-turbinate nasal swab from both nostrils, perform and interpret the Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test. All procedures for testing and result interpretation, including sample collection and extraction will be conducted by the lay user following the Instructions for Use provided in the kit.
  The first NP swab sample will be used to conduct a Panbio™ COVID- 19/FluA&B Rapid Panel Professional Use test.
  The second NP swab sample will be eluted in Universal Transport Medium (UTM) provided by Abbott/the Core Laboratory, labelled and stored, according to the laboratory manual. UTM samples will be shipped to the Core Laboratory for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2, according to the laboratory manual.
  Interventions: Diagnostic Test: Panbio™

INTERVENTIONS:
Diagnostic Test: Panbio™ — The Panbio™ COVID-19/Flu A&B Rapid Panel Professional use device is a visual lateral flow assay, for rapid immunochromatographic qualitative detection of COVID-19 antigen, Influenza A antigen and Influenza B antigen in nasopharyngeal swabs, collected by a trained health worker.
  The Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test device is a visual lateral flow assay, for rapid immunochromatographic qualitative detection of COVID-19 antigen, Influenza A antigen and Influenza B antigen in self-collected mid-turbinate nasal swabs. The test is designed to be used by lay users
  Other Names: Panbio™ COVID-19/Flu A&B Rapid Panel Professional Use Product; Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test Device

SUMMARY:
This study is designed as an international prospective, multicentric, clinical study to investigate the performance and usability of the Panbio™ COVID-19/Flu A&B Rapid Panel Professional Use and Self- Test devices for the qualitative detection of COVID-19 antigen, Influenza A antigen and Influenza B antigen in human nasopharyngeal (NP) and mid-turbinate nasal swabs, respectively.

This study is part of the performance evaluation to support the CE conformity assessment procedures.

DETAILED DESCRIPTION:
In total, a minimum of 1531 male and female subjects will be prospectively enrolled at multiple clinical sites. A minimum of 100 lay users will also be asked to interpret randomly assigned mock devices.

After obtaining written informed consent, a study-specific subject identification number (ID) will be assigned to the subject. All eligible subjects will be assigned to both Professional Use arm and the Self-Test arm of the study. Subject demographics and a brief medical history will be collected.

Lay users (self-tester or caregiver) will first collect one mid-turbinate nasal swab from both nostrils, and perform and interpret the Panbio™ Rapid Panel ST device, under the observation of a trained observer. All procedures for testing and result interpretation, including sample collection and extraction, will be conducted following the IFU provided in the kit. Each Panbio™ Rapid Panel ST result will be interpreted firstly by the lay user and followed immediately by the observer who will also photograph the test at the time of interpretation. Each lay user will fill out a user evaluation questionnaire, and a study staff member will complete an observer questionnaire for each lay user. A minimum of 100 lay users will also read mock device tests presented by a study staff member. Mock devices (simulated to represent testing results) will be used for usability testing (result interpretation).

A study staff member will then collect two NP swabs (one swab from each nostril) from all subjects. The first NP swab sample will be used to conduct a Panbio™ Rapid Panel PU test, following the IFU. The test result will be photographed at the time of result interpretation. Each study staff member who performs a Panbio™ Rapid Panel PU test will fill out a user evaluation questionnaire once, to assess the usability of the device.

The second NP swab sample will be eluted in Universal Transport Medium (UTM) provided by Abbott/the Core Laboratory, labelled and stored, according to the laboratory manual. UTM samples will be shipped to the Core Laboratory for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2, according to the laboratory manual.

Each subject's demographic information, education, symptomology data, test results and questionnaires, where relevant, will be recorded on source documentation and transferred to an Electronic Data Capture system.

ELIGIBILITY:
Inclusion Criteria:

Subjects from all age groups, able and willing to provide written informed consent or assent, suspected of having a respiratory viral infection consistent with COVID-19 and/or Flu by their healthcare provider within the first five days of the onset of symptoms, and presenting at least two of the following symptoms: fever, headache, tiredness, dry cough, sore throat, runny or stuffy nose, muscle aches, loss of smell, loss of taste or shortness of breath, will be prospectively enrolled.

Exclusion Criteria:

* Subject has had a nasal or a NP swab taken within the last 4 hours and is not available for further testing after 4 hours has elapsed.
* Subject has active nose bleeds or acute facial injuries/trauma.
* Subject has received a nasal vaccine (i.e., FluMist®) within the previous fourteen (14) days.
* Subject is currently taking or has taken an antiviral medication- e.g., Amantadine, Rimantadine, Relenza® (Zanamivir), Tamiflu® (Oseltamivir Phosphate), and Flumadine®-for influenza or COVID-19 within the previous thirty (30) days.
* Subject is currently enrolled in a study to evaluate an investigational drug.
* Self-tester or caregiver has prior medical or laboratory training.
* Self-tester or caregiver has a visual impairment that cannot be restored using glasses or contact lenses or lay user is unable to read the Instructions for Use.
* Subject has a condition deemed unfit to safely perform the test.
* Subject is unwilling or unable to provide informed consent.
* Vulnerable populations as deemed inappropriate for the study by the site's PI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the Panbio™ COVID-19/Flu A&B Rapid Panel device. | "up to 24 months"
  To assess the clinical performance (sensitivity/specificity) of the Panbio™ COVID-19/Flu A&B Rapid Panel in fresh collected mid-turbinate nasal swab specimens from individuals suspected of respiratory viral infection consistent with COVID-19 and/or Flu by their healthcare provider within the first five days of the onset of symptoms in a Near Patient Testing setting, compared to Flu and SARS-CoV-2 RT-PCR tested using NP swab samples. Concordance analyisis of investigational device and reference method. Acceptance criterion: Sensitivity >80%, Specificity >95%
  To assess the clinical performance (sensitivity/specificity) of the Panbio™ COVID- 19/Flu A&B Rapid Panel Self-Test device, as performed by lay users (self-testers or caregivers) using fresh collected mid-turbinate nasal self- collected samples, when compared to Flu and SARS-CoV-2 RT- PCR using NP swab samples.

SECONDARY OUTCOMES:
Concordance of self-test and professional use device | "up to 24 months"
  To assess concordance between the Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test device using mid-turbinate nasal self-collected samples and the Professional Use device using NP samples collected by a trained health worker.
Usability of the professional use device | "up to 24 months"
  To assess the usability of the Panbio™ COVID-19/Flu A&B Rapid Panel professional use device when used by trained healthcare workers. Usability is assessed by a questionnaire.
Usability of the self test device | "up to 24 months"
  To assess the usability of the Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test device, as performed by lay users with no laboratory or clinical experience. Usability testing will also comprise of the interpretation of mock devices. User and observer questionnaires will also be utilized to assess usability.

CONTACTS AND LOCATIONS:
Locations (1):
- UCCT @ AFC Urgent Care- Easley, Easley, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No